CLINICAL TRIAL: NCT03531086
Title: Exploring Dopamine Transporter Single-photon Emission Computer Tomography Quantification as a Measure of Disease Progression in Idiopathic Parkinson's Disease
Brief Title: Idiopathic Parkinson's Progression and Dopamine Transporter SPECT
Status: Completed | Type: Observational
Sponsor: Julie Gurwell (Other)
Responsible Party: Sponsor-Investigator, Julie Gurwell, Associate Professor Director of Advanced Practice Providers, Neurology, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 42475
Record Dates: First submitted 2018-05-08; First posted 2018-05-21 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Parkinson Disease
Keywords: dopamine transporter binding
MeSH Terms: conditions — Parkinson Disease | interventions — ioflupane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ioflupane I123: Participants will receive Ioflupane I123 as an adjunct diagnostic tool in combination with single photon emission computer tomography (SPECT) to evaluate striatal dopamine transporter. Patients will serve as their own control longitudinally.
  Interventions: Drug: Ioflupane I 123

INTERVENTIONS:
Drug: Ioflupane I 123 — Ioflupane I 123 will be administered IV push prior to SPECT imaging
  Other Names: DaTscan

SUMMARY:
DaTscanTM Ioflupane I123, a radiopharmaceutical will be used as an adjunct diagnostic tool in combination with single photon emission computed tomography (SPECT) to evaluate striatal dopamine transporter (DAT) distribution in patients with idiopathic Parkinson's disease. Patients will be monitored twice - once at baseline, and again after 1 year - to identify potential biomarkers for progression of Parkinson's disease.

DETAILED DESCRIPTION:
Background: Idiopathic Parkinson's disease (PD) is a neurodegenerative disorder involving loss of dopaminergic neurons in the substantia nigra and subsequent dysfunction in the striatum. The diagnosis of PD remains a clinical diagnosis based on patient history and physical exam findings. In 2011 the FDA approved the use of DaTscanTM Ioflupane I123, a radiopharmaceutical to be used as an adjunct diagnostic tool in combination with single photon emission computed tomography (SPECT) to evaluate striatal dopamine transporter (DAT) distribution in patients with an unclear diagnosis of parkinsonism vs essential tremor (Bajaj et al., 2013). Because the loss of DAT binding in the striatum reflects the loss of dopaminergic neurons in parkinsonism, DAT SPECT is considered a highly sensitive test for these disorders (Ba and Martin, 2015). The major clinical uncertainty with DAT SPECT imaging is whether or not quantitative analysis can be utilized to determine progressive degeneration over time and serve as a quantitative biomarker for changes in striatal dopaminergic integrity in correlation with clinical worsening in patients with idiopathic PD. In 3 small studies using two other ligands, 18F-dopa and I123β-CIT, striatal uptake declined annually by 12.5-13%, and 2.4% - 7.1%, respectively (Morrish et al., 1996; Nurmi et al., 2000; Pirker et al., 2012). Current analytical methodologies have focused on establishing differences between the PD and control groups, but have not explored the technology for tracking disease progression with Ioflupane I123, using the patient as their own control. The goal of this proposed study is to evaluate the validity of quantitative measurements in DAT SPECT scans in determining disease progression in subjects with idiopathic PD. Data from this pilot study would contribute significantly to future applications for investigating translational research strategies to restore dopaminergic cell function in PD. More specifically, the ability of autologous peripheral nerve grafts, acting as a source of neuroregenerative growth factors, is being investigated in PD subjects undergoing deep brain stimulation (Craig van Horne, PI). As there are no current biomarkers for PD progression, it is critical to evaluate the potential for DAT SPECT to serve as an analytical tool for the quantification of dopaminergic functional integrity. This study is designed to test the ability of DAT SPECT to be used as an effective methodology for tracking disease progression where patients serve as their own control.

Objectives: The specific aim is to evaluate the ability of DAT SPECT quantification to track disease progression in subjects with idiopathic Parkinson's disease by comparing baseline scans to those obtained 12 months later. The quantified DAT SPECT data will be clinically correlated to the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) motor scores and Hoehn and Yahr stage obtained at baseline and at 12 months.

Study Design: This will be an initial phase of a prospective study evaluating DAT SPECT quantification in subjects with idiopathic Parkinson's disease. The clinical severity of PD will be measured by MDS-UPDRS motor scores and the Hoehn and Yahr scale. Data will be acquired at baseline, and 12 months. The subject will serve as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40-75
* Able to give informed consent
* Show a positive response to carbidopa/levodopa
* Hoehn and Yahr score 1-3

Exclusion Criteria:

* Under the age of 40 or over the age of 75
* Unable to give informed consent
* Nonresponsive to carbidopa/levodopa
* Hoehn and Yahr score 4-5
* Unable to discontinue medications which might interfere with DaTscan TM imaging
* Inability to lie still for 30-45 minutes during CT-SPECT imaging
* Pregnancy or Nursing
* Severe kidney function impairment
* Unable to tolerate iodine containing products
* Patients with deep brain stimulation (DBS) or a history of any other brain surgery

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects to be recruited during office visits at the University of Kentucky.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in dopamine transporter binding in idiopathic Parkinson's Disease progression. | 1-year
  Patients will receive dopamine transporter SPECT imaging at baseline and after one year to investigate the ability of this technique to quantitatively assess neurodegeneration in the substantia nigra.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gurwell, PhD, PA-C, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Department of Neurology, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share data.